CLINICAL TRIAL: NCT05307575
Title: Cognition, Emotion/Behavior, Functionality and Brain Connectivity in Recovered COVID-19 Patients
Brief Title: Neurobehavior and Brain Connectivity in Post COVID-19 Patients
Acronym: NAUTILUS
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: University of Barcelona (Other); Universitat Politècnica de Catalunya (Other)
Responsible Party: Principal Investigator, Maite Garolera, Chief of the Neuropsychology Unit and Director of the Brain, Cognition, and Behavior Research Group (C3-CST) of CST., Consorci Sanitari de Terrassa
Other Study IDs: 202111-30-31-32 Fundació La Ma
Record Dates: First submitted 2022-03-31; First posted 2022-04-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post-COVID Syndrome
Keywords: COVID-10; Cognition; Mental Health; Neuroimage; Machine Learning
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post-COVID syndrome (PCS) Severe COVID-19: Severe COVID-19 with PCS with cognitive complains
- Post-COVID syndrome (PCS) Mild COVID-19: Mild COVID-19 with PCS with cognitive complains
- Controls: Healthy adult controls

SUMMARY:
COVID-19 neurological effects can generate long-term neurobehavioral dysfunction. Our main objective is to examine the impact of COVID-19 on neurobehavior and its relationship with illness severity. Besides, we aim to study structural and functional brain connectivity in a subsample of middle-aged post-COVID-19 individuals. Finally, we aim to develop predictive models of neurobehavioural evolution in post-COVID-19 based on multimodal data.

DETAILED DESCRIPTION:
NAUTILUS is an observational, cross-sectional, and multicenter study. It will be performed at 22 public hospitals. Two groups of COVID-19 adults (Severe N=210, Moderate-mild N=210, WHO criteria) reporting cognitive complaints will compare to healthy controls (N=210). They will be assessed on neurobehavioral status. We will perform brain MRI in a subsample (N=120, 40 per group), and we will obtain potential biomarkers of neural damage (smell function, retinal blood plexuses integrity, and inflammation). Moreover, we will use machine learning-based algorithms based on demographics, previous pathologies, lifestyle, clinical data, and biomarkers to predict neurobehavioral models.

Expected results: Identify the neurobehavioral impact of post-COVID-19 individuals and the discriminative power of multimodal biomarkers in adverse outcomes. Our result would help develop clinically useful models to predict the neurobehavioral impact to develop future personalized and preventive intervention strategies.

ELIGIBILITY:
PCS from SEVERE COVID-19 group

Inclusion Criteria:

* Confirmed diagnosis of COVID-19 according to WHO interim with signs and symptoms of the severe disease during the acute phase
* Presence of cognitive complaints after COVID-19 diagnosis
* Participants have to be discharged from the hospital at least three months before inclusion
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki

Exclusion Criteria:

* Participants have symptoms of delirium according to Delirium Rating Scale-revised 98
* Established diagnosis before COVID-19 disease of psychiatric, neurological, neurodevelopmental disorder or systemic pathologies are known to cause cognitive deficits
* Motor or sensory alterations that impede the neuropsychological examination
* Participants with a metal prosthesis (for MRI studies)
* Subjects suffering from claustrophobia or requiring sedation due to high anxiety (for MRI studies)

PCS from MILD COVID-19 group

* Confirmed diagnosis of MILD COVID-19 according to WHO interim
* Presence of cognitive complaints after COVID-19 diagnosis
* Participants have to be diagnosed with COVID-19 at least three months before inclusion
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki

Exclusion Criteria:

* Established diagnosis before COVID-19 disease of psychiatric, neurological, neurodevelopmental disorder or systemic pathologies are known to cause cognitive deficits
* Motor or sensory alterations that impede the neuropsychological examination
* Participants with a metal prosthesis (for MRI studies)
* Subjects suffering from claustrophobia or requiring sedation due to high anxiety (for MRI studies)

Healthy adult CONTROL group

Inclusion Criteria:

* Healthy people who have not had COVID-19
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki

Exclusion Criteria:

* the same as COVID-19 groups

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PCS from severe and mild COVID-19 group will be recruited in hospital and primary care services.
  The control population will be searched in the general population through primary care centers, the media, social networks, and they will be offered to participate in the study without remuneration.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Differences between groups in auditory attention | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Auditory attention is measured with Digit Span Forward. Participants are asked to repeat numbers in the same order as read aloud by the examiner. Higher scores mean a better outcome.
Differences between groups in working memory | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Working memory is measured with Digit Span Backward. Participants are asked to repeat the numbers in the reverse order of that presented by the examiner. Higher scores mean a better outcome.
Differences between groups in language | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Language is measured with the Boston Naming Test. It consists of 60 line drawings of objects of graded difficulty, ranging from very common things to less familiar objects. The total score is the sum of correct answers. Higher scores mean a better outcome.
Differences between groups in verbal memory | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Verbal memory is measured with the Auditory Verbal Learning Test (AVLT). It is a word-learning test where five presentations of a 15-word list are given, each followed by an attempted recall. This is followed by a second 15-word interference list (list B), followed by recall of list A. Delayed recall and recognition are also tested. Higher scores mean a better outcome.
Differences between groups in visual memory | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Visual memory is measured with the Rey-Osterrieth Complex Figure (ROCF) test. The participants are asked to copy complex geometric shapes and then reproduce them from memory. A delayed recall is also tested. Higher scores mean a better outcome.
Differences between groups in psychomotor speed | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Processing speed is measured with Coding subtest of WAIS. Participants are asked to use a key to put in the appropriate symbols for a list of numbers. Higher scores mean a better outcome.
Differences between groups in perceptual reasoning | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Perceptual reasoning is measured with Matrix reasoning subtest of WAIS. Participants are asked to choose which of some possible options the missing picture is from matrix of abstract pictures. Higher scores mean a better outcome.
Differences between groups in executive function | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  A composite score is made with the z-scores of phonemic (sum of the three letters) and semantic fluency, Trail Making Test B (time) and STROOP test (color-word interference total items in 120 seconds).
Differences between groups in social cognition | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Social cognition is measured with the Reading the Mind in the Eyes Test. Participants are asked to choose the emotional state that best describes the eyes, choosing between one of four possible emotions in the 36 photographs of male and female eyes depicting emotional states. Higher scores mean a better outcome.
Differences between groups in anxiety | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Anxiety is measured with the 7-item Generalized Anxiety Disorder Scale (GAD-7), a Likert-type scale with questions ranging from "not at all" (0 points) to "nearly every day" (3 points). The maximum score is 24. Higher scores mean a worse outcome.
Differences between groups in depression | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Depression is measured with the Patient Health Questionnaire-9 (PHQ-9) which scores each of the 9 DSM-IV criteria as "not at all" (0 points) to "nearly every day" (3 points). Higher scores mean a worse outcome.
Differences between groups in Post-traumatic Stress Disorder | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Post-Traumatic Stress Disorder is measured with The Post-Traumatic Stress Disorder Checklist (PCL-5), a 20-item questionnaire corresponding to the DSM-5 symptom criteria for PTSD, which scores each criterion as "not at all" (0 points) to "extremely" (4 points). The ratings of items are added together to calculate the total score (range=0-80). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Differences between groups in Fatigue | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Fatigue is measured with the Chalder Fatigue Scale, an 11-item questionnaire measuring the severity of physical and mental fatigue on two separate subscales. Seven items represent physical fatigue (items 1-7) and 4 represent mental fatigue (items 8-11). Each item " less than usual" (0) to " much more than usual" (3). The ratings of items are added together to calculate the total score (range=0-33). High scores represent high levels of fatigue.
Differences between groups in Quality of Life | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Quality of life is measured with a 12-item World Health Organization Disability Assessment Schedule-II (WHODAS-II). Patients are asked to state the level of difficulty experienced, considering how they usually do the activity. The scale scores each item as "none" (1) to "cannot do" (5). The total score is calculated with an SPSS syntax, and the range varies from 0 to 100, with higher scores reflecting more significant disability.
Differences between groups in White Matter integrity | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  White matter integrity: tractography measured by MRI
Differences between groups in brain Volumetry | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Grey and white matter volume measured by MRI
Differences between groups in Resting-state connectivity | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Resting state brain activity using fMRI
Differences between groups in plasmatic Interleukin- 6 (IL-6) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of IL-6 are measured with enzyme-linked immunosorbent assay (ELISA) Kit
Differences between groups in plasmatic Nerve Growth Factor (NGF) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of NGF are measured with ELISA Kit
Differences between groups in plasmatic Glial Fibrillary Acidic Protein (GFAp) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of GFAp are measured with ELISA Kit
Differences between groups in plasmatic lipid peroxidation products | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of malondialdehyde are measured with TBARS assay method
Differences between groups in plasmatic Ferritin | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of Ferritin are measured with biochemical assay
Differences between groups in plasmatic C-Reactive Protein (CRP) | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  The plasma levels of CRP are measured with high sensitivity c-reactive protein ELISA Kit
Differences between groups in smell function | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Smell function is evaluated with the University of Pennsylvania Smell Identification Test (UPSIT), which measures the individual's ability to detect odors at a suprathreshold level. The UPSIT comprises four booklets, each of which contains ten pages. An odorized "scratch & sniff" label is present on each booklet page. The subject scratches the label and then indicates which of the four response alternatives best matches the perceived smell. A score ranging from 6-18 means anosmia, 19-25 means severe microsmia, 26-30 in women and 26-29 in men means moderate microsmia, 31-34 in women and 30-33 in men means mild microsmia and a score of more than 34 in women and 33 in men means normosmia.
Differences between groups retinal plexuses integrity | At the time of inclusion of the participant, between 3 and 12 months from the start of COVID-19
  Retinal plexuses integrity is measured with Optical Coherence Tomography Angiography (OCTA)

CONTACTS AND LOCATIONS:
Overall Officials: Maite Garolera, PhD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carreras-Vidal L, Pacheco-Jaime L, Ariza M, Cano N, Garolera M, Garcia-Vicente C, Roura I, Capdevila-Lacasa C, Oltra J, Pardo J, Martin-Barcelo C, Campabadal A, Sala-Llonch R, Bargallo N, Barrue C, Bejar J, Cortes CU, Junque C; NAUTILUS-Project Collaborative Group; Segura B. Functional brain abnormalities in post COVID-19 condition and their relationship with cognition. Sci Rep. 2025 Jul 1;15(1):22259. doi: 10.1038/s41598-025-00739-3. PMID 40595626
- [Derived] Pacheco-Jaime L, Garcia-Vicente C, Ariza M, Cano N, Garolera M, Carreras-Vidal L, Roura I, Capdevila-Lacasa C, Oltra J, Pardo J, Martin-Barcelo C, Campabadal A, Sala-Llonch R, Bargallo N, Barrue C, Bejar J, Cortes CU, Junque C, Segura B; NAUTILUS-Project Collaborative Group. Structural brain changes in post-COVID condition and its relationship with cognitive impairment. Brain Commun. 2025 Feb 12;7(1):fcaf070. doi: 10.1093/braincomms/fcaf070. eCollection 2025. PMID 40008326
- [Derived] Ariza M, Bejar J, Barrue C, Cano N, Segura B; NAUTILUS Project Collaborative Group; Cortes CU, Junque C, Garolera M. Cognitive reserve, depressive symptoms, obesity, and change in employment status predict mental processing speed and executive function after COVID-19. Eur Arch Psychiatry Clin Neurosci. 2025 Jun;275(4):973-989. doi: 10.1007/s00406-023-01748-x. Epub 2024 Jan 29. PMID 38285245
- [Derived] Ariza M, Cano N, Segura B, Adan A, Bargallo N, Caldu X, Campabadal A, Jurado MA, Mataro M, Pueyo R, Sala-Llonch R, Barrue C, Bejar J, Cortes CU; NAUTILUS Project Collaborative Group; Garolera M, Junque C. COVID-19 severity is related to poor executive function in people with post-COVID conditions. J Neurol. 2023 May;270(5):2392-2408. doi: 10.1007/s00415-023-11587-4. Epub 2023 Mar 20. PMID 36939932
- [Derived] Ariza M, Cano N, Segura B, Adan A, Bargallo N, Caldu X, Campabadal A, Jurado MA, Mataro M, Pueyo R, Sala-Llonch R, Barrue C, Bejar J, Cortes CU; NAUTILUS-Project Collaborative Group; Junque C, Garolera M. Neuropsychological impairment in post-COVID condition individuals with and without cognitive complaints. Front Aging Neurosci. 2022 Oct 20;14:1029842. doi: 10.3389/fnagi.2022.1029842. eCollection 2022. PMID 36337708